CLINICAL TRIAL: NCT01436305
Title: Optimization of NULOJIX® (Belatacept) Usage as a Means of Avoiding CNI and Steroids in Renal Transplantation (CTOT-10)
Brief Title: Optimization of NULOJIX® Usage As A Means of Avoiding CNI and Steroids in Renal Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Secondary to safety concerns plus change in Campath® (alemtuzumab) availability.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CTOT-10
Record Dates: First submitted 2011-09-13; First posted 2011-09-19 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-08

CONDITIONS: Kidney Transplantation; Renal Transplantation
Keywords: immunosuppressive (IS) regimens; long-term graft function; CNI (calcineurin Inhibitor )-free IS regimen; CNI (calcineurin Inhibitor ) IS regimen; corticosteroids
MeSH Terms: interventions — Alemtuzumab; Mycophenolic Acid; Basiliximab; Tacrolimus; Abatacept; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tac maintenance (Active Comparator): Group 1 Study Therapy Regimen:Induction with alemtuzumab and maintenance immunosuppression with tacrolimus and mycophenolate mofetil (MMF).
  Campath® (alemtuzumab); long-term Prograf® (tacrolimus), or equivalent ; CellCept® (mycophenolate mofetil- MMF), or equivalent , and 4 day course of MEDROL® (methylprednisolone)
  Interventions: Drug: Alemtuzumab; Drug: MMF; Drug: tacrolimus; Drug: methylprednisolone
- Belatacept maintenance (Experimental): Group 2 Study Therapy Regimen: Induction with alemtuzumab and maintenance with Nulojix® (belatacept) and mycophenolate mofetil (MMF).
  Campath® (alemtuzumab); Nulojix® (belatacept); CellCept® (mycophenolate mofetil- MMF), or equivalent, and 4 day course of MEDROL®(Methylprednisolone)
  Interventions: Drug: Alemtuzumab; Drug: MMF; Biological: Belatacept; Drug: methylprednisolone
- Basiliximab induction/Short-term Tac (Experimental): Short term = 3 months
  Group 3 Study Therapy Regimen: Induction with 2 doses of basiliximab and tacrolimus for 84 days and maintenance with Nulojix® (belatacept) and mycophenolate mofetil (MMF).
  Simulect® (basiliximab); Nulojix® (belatacept); short-term course of Prograf® (tacrolimus), or equivalent; CellCept® (mycophenolate mofetil- MMF), or equivalent, and 4 day course of MEDROL® (methylprednisolone)
  Interventions: Drug: MMF; Biological: Basiliximab; Drug: Short-term Tac; Biological: Belatacept; Drug: methylprednisolone

INTERVENTIONS:
Drug: Alemtuzumab — Induction therapy. Group 1 and 2 study therapy regimens include induction with alemtuzumab, administered as a single intravenous dose intra-operatively over a period of 2 hours.
  Other Names: Campath®
  Arms: Belatacept maintenance; Tac maintenance
Drug: MMF — All treatment groups (e.g., Group 1, 2 and 3): Administered at a target dose of 1000 mg by mouth twice daily beginning on the day of surgery or post operative day 1 and adjusted as clinically warranted.
  Note: Myfortic® (mycophenolate sodium) may be used as a replacement for MMF, at a dose of 720 mg taken by mouth twice daily.
  Other Names: mycophenolate mofetil; CellCept®
Biological: Basiliximab — Induction therapy. Group 3 study therapy regimen includes induction with basiliximab, administered in two doses: 1 dose administered within 2 hours prior to transplantation surgery and the 2nd dose 4 days after transplantation (unless held due to contraindication[s])
  Other Names: Simulect®
  Arms: Basiliximab induction/Short-term Tac
Drug: Short-term Tac — Short-term (3 months)
  Other Names: tacrolimus; Prograf®
  Arms: Basiliximab induction/Short-term Tac
Drug: tacrolimus — maintenance
  Other Names: Prograf®
  Arms: Tac maintenance
Biological: Belatacept — maintenance
  Other Names: Nulojix®
  Arms: Basiliximab induction/Short-term Tac; Belatacept maintenance
Drug: methylprednisolone — All study treatment groups: administration started on the day of transplant and tapered over a 4 day course.
  Other Names: MEDROL®

SUMMARY:
The purpose of this study was to assess whether a new drug, Nulojix® (belatacept), would minimize serious long term side effects associated with anti-rejection medications while still protecting the new kidney from damage. The researchers also wanted to learn more about the safety of this treatment and long term health of the transplanted kidney.

DETAILED DESCRIPTION:
Dialysis or kidney transplant are the two ways to treat kidney failure. Transplant recipients have to take anti-rejection medications to prevent their immune system (the body's natural defense system against illness) from rejecting their new kidney. Most patients who undergo a kidney transplant must take these anti-rejection medications for the rest of their lives. Taking standard anti-rejection medications for a long time can cause serious side effects, including kidney damage. There would be a benefit to finding new anti-rejection medications that work just as well, but don't damage the kidney.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, 18-65 years of age at the time of enrollment;
* Ability to understand and provide written informed consent;
* Candidate for primary renal allograft from either a living or deceased-donor;
* No known contraindications to study therapy using NULOJIX® (belatacept);
* Female participants of childbearing potential must have a negative pregnancy test upon study entry;
* Female and male participants with reproductive potential must agree to use FDA approved methods of birth control during participation in the study and for 4 months following completion of the study;
* Flow-based PRA within last 12 months (in absence of a sensitizing event) of < 30% as determined by each participating study center. If the subject experienced a sensitizing event after the PRA test date, then the PRA must be repeated and confirmed <30%;
* Negative crossmatch or a PRA of 0% on historic and admission sera as determined by each participating study center.
* A documented negative TB test within the 12 months prior to transplant. If documentation is not present at the time of transplantation, and the subject does not have any risk factors for TB, a TB-specific interferon gamma release assay (IGRA) may be performed.

Exclusion Criteria:

* Need for multi-organ transplant;
* Recipient of previous organ transplant;
* EBV sero-negative (or unknown) recipients;
* Active infection including hepatitis B, hepatitis C, or HIV;
* Individuals who have required treatment with prednisone or other immunosuppressive drugs within 1 year prior to transplant;
* Individuals undergoing transplant using organs from extended criteria donor (ECD) or donation after cardiac death (DCD) donors;
* HLA identical living donors;
* Individuals at significant risk of early recurrence of the primary renal disease including FSGS and MPGN type 2 or any other disease that in the opinion of the investigator is at increased likelihood of recurrence and which may result in rapid decline in renal function;
* Individuals previously treated with NULOJIX® (belatacept);
* Any condition that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements;
* Use of investigational drugs within 4 weeks of enrollment;
* Known hypersensitivity to mycophenolate mofetil (MMF) or any of the drug's components;
* Administration of live attenuated vaccine(s) within 8 weeks of enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Newell, MD, PhD, Study Chair — Emory University; Christian P. Larsen, MD, DPhil, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia

REFERENCES:
- [Result] Newell KA, Mehta AK, Larsen CP, Stock PG, Farris AB, Mehta SG, Ikle D, Armstrong B, Morrison Y, Bridges N, Robien M, Mannon RB. Lessons Learned: Early Termination of a Randomized Trial of Calcineurin Inhibitor and Corticosteroid Avoidance Using Belatacept. Am J Transplant. 2017 Oct;17(10):2712-2719. doi: 10.1111/ajt.14377. Epub 2017 Jul 3. PMID 28556519
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Clinical Trials in Organ Transplantation (CTOT) website — https://www.ctotstudies.org/index.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three sites in the United States enrolled a total of 19 participants in the study.
Groups:
- Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus: Induction: Alemtuzumab was administered in a single intravenous dose of 30 mg intra-operatively over a period of 2 hours.
  Maintenance: Starting on the day of surgery or post-operative day one, participants underwent maintenance therapy.
  Mycophenolate mofetil (MMF) was given at a dose of 1000 mg by mouth twice a day of which was adjusted as clinically warranted. Mycophenolate sodium could be used to replace MMF at a dose 720 mg by mouth twice a day.
  Methylprednisone was administered at a dose of 500 mg on the day of transplant, and tapered to 250 mg day 1 post-transplant, 125 mg day 2 post-transplant, 60 mg day 3 post-transplant, 30 mg day 4 post-transplant.
  Tacrolimus was given at a dose of 0.1 mg/kg twice a day by mouth, which was adjusted to target trough levels of 8-12 ng/ml during the first 24 weeks post-transplant, then adjusted to target trough levels of 5-8 ng/ml thereafter.
- Induction: Alemtuzumab, Maintenance: MMF + Belatacept: Induction: Alemtuzumab was administered in a single intravenous dose of 30 mg intra-operatively over a period of 2 hours.
  Maintenance: Starting on the day of surgery or post-operative day one, participants underwent maintenance therapy.
  Mycophenolate mofetil (MMF) was given at a dose of 1000 mg by mouth twice a day of which was adjusted as clinically warranted. Mycophenolate sodium could be used to replace MMF at a dose 720 mg by mouth twice a day.
  Methylprednisone was administered at a dose of 500 mg on the day of transplant, and tapered to 250 mg day 1 post-transplant, 125 mg day 2 post-transplant, 60 mg day 3 post-transplant, 30 mg day 4 post-transplant.
  Belatacept was given at a dose of 10 mg/kg on Day 0, then at days 4, 14, 28, 56 and 84. After Day 84, participants received 5 mg/kg every 4 weeks.
- Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac: Induction: Basiliximab was administered in 2 doses of 20 mg each, 2 hours prior to surgery and 4 days post-transplantation.
  Maintenance: Starting on the day of surgery or post-operative day one, participants underwent maintenance therapy.
  Mycophenolate mofetil (MMF) was given at a dose of 1000 mg by mouth twice a day of which was adjusted as clinically warranted. Mycophenolate sodium could be used to replace MMF at a dose 720 mg by mouth twice a day.
  Methylprednisone was given at a dose of 500 mg on Day 0, and tapered to 250 mg day 1 post-transplant, 125 mg day 2 post-transplant, 60 mg day 3 post-transplant, 30 mg day 4 post-transplant.
  Belatacept was given at a dose of 10 mg/kg on Day 0, then at days 4, 14, 28, 56 and 84. After Day 84, participants received 5 mg/kg every 4 weeks.
  Tacrolimus was given at a dose of 0.1 mg/kg twice a day by mouth, then adjusted to target trough levels: 8-12 ng/ml by Day 29, 5-8 ng/ml by Day 57, 3-5 ng/ml by Day 85 then stopped.
Period: Overall Study
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Started | 6 | 6 | 7
Completed | 4 | 2 | 7
Not Completed | 2 | 4 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac | Total
Number analyzed (Participants) | 6 | 6 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (13.1) | 43.3 (9.5) | 49.1 (9.0) | 46.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 6
  Male | 4 | 3 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 4 | 16
  Unknown or Not Reported | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 5 | 8
  White | 4 | 4 | 2 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 7 | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Glomerular Filtration Rate (GFR) Calculated for Each Treatment Group Using the CKD-EPI Equation at Wk 52
Description: GFR was calculated using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI). A score of ≥ 90 means kidney function is normal. A score between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease. Scores between 30 and 59 indicates moderately reduced kidney function. Scores between 15 and 29 indicate severely reduced kidney function. Scores below 15 indicate very severe or endstage kidney failure.
Time Frame: Week 52
Population: Intent-to-treat population with measurable data at Week 52
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 4 | 3 | 7
mL/min/1.73m^2 | 55.9 (8.9) | 51.6 (23.5) | 58.3 (12.2)

2. Secondary Outcome: Count of Participants With Biopsy Proven Acute Rejection at Any Time Post-Transplant
Description: Biopsy proven acute rejection was defined as histologic evidence of borderline or higher cellular rejection per local pathologist.
Time Frame: Transplantation through last study visit (up to week 156)
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Participants | 3 | 2 | 5

3. Secondary Outcome: Count of Participants With Estimated Glomerular Filtration Rate (GFR) < 60 mL/Min/1.73 m^2 by CKD EPI
Description: GFR was calculated using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI). A score of ≥90 means kidney function is normal. A score between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease. Scores between 30 and 59 indicates moderately reduced kidney function. Scores between 15 and 29 indicate severely reduced kidney function. Scores below 15 indicate very severe or endstage kidney failure. This measure specifically looked at participants with scores less than 60.
Time Frame: Week 52, Week 104, and Week 156
Population: Intent-to-treat population with available data at Weeks 52, 104 and 156.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 4 | 3 | 7
Participants
  Week 52 | 3 | 2 | 4
  Week 104: number analyzed (Participants) | 3 | 2 | 7
  Week 104 | 2 | 1 | 3
  Week 156: number analyzed (Participants) | 3 | 2 | 7
  Week 156 | 2 | 1 | 2

4. Secondary Outcome: Count of Participants by Chronic Kidney Disease (CKD) Stage Post-Transplant
Description: The stages of Chronic Kidney Disease are defined using the participant's GFR value as indicated below:
  Stage 1 if GFR value is ≥90; Stage 2 if GFR value is ≥60 and < 90; Stage 3A if 45 ≤GFR < 60; Stage 3B if 30 ≤ GFR < 45; Stage 4 if 15 ≤GFR < 30;l Stage 5 if GFR < 15.
  Stage 1 means kidney function is normal. Stage 2 indicates mildly reduced kidney function, pointing to kidney disease. Stages 3A and 3B indicate moderately reduced kidney function. Stage 4 indicates severely reduced kidney function. Stage 5 indicates very severe or end stage kidney failure.
Time Frame: Week 52, Week 104, and Week 156
Population: Intent-to-treat population with available data at Weeks 52, 104 and 156
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 4 | 3 | 7
Participants
  Week 52 - Stage 1 | 0 | 0 | 0
  Week 52 - Stage 2 | 1 | 1 | 3
  Week 52 - Stage 3A | 3 | 1 | 3
  Week 52 - Stage 3B | 0 | 0 | 1
  Week 52 - Stage 4 | 0 | 1 | 0
  Week 104 - Stage 1: number analyzed (Participants) | 3 | 2 | 7
  Week 104 - Stage 1 | 0 | 1 | 1
  Week 104 - Stage 2: number analyzed (Participants) | 3 | 2 | 7
  Week 104 - Stage 2 | 1 | 0 | 3
  Week 104 - Stage 3A: number analyzed (Participants) | 3 | 2 | 7
  Week 104 - Stage 3A | 1 | 1 | 2
  Week 104 - Stage 3B: number analyzed (Participants) | 3 | 2 | 7
  Week 104 - Stage 3B | 1 | 0 | 1
  Week 104 - Stage 4: number analyzed (Participants) | 3 | 2 | 7
  Week 104 - Stage 4 | 0 | 0 | 0
  Week 156 - Stage 1: number analyzed (Participants) | 3 | 2 | 7
  Week 156 - Stage 1 | 0 | 0 | 0
  Week 156 - Stage 2: number analyzed (Participants) | 3 | 2 | 7
  Week 156 - Stage 2 | 1 | 1 | 5
  Week 156 - Stage 3A: number analyzed (Participants) | 3 | 2 | 7
  Week 156 - Stage 3A | 1 | 1 | 1
  Week 156 - Stage 3B: number analyzed (Participants) | 3 | 2 | 7
  Week 156 - Stage 3B | 1 | 0 | 1
  Week 156 - Stage 4: number analyzed (Participants) | 3 | 2 | 7
  Week 156 - Stage 4 | 0 | 0 | 0

5. Secondary Outcome: Count of Participants With CKD Stage 4 or 5
Description: The stages of Chronic Kidney Disease are defined using the participant's GFR value as indicated below.
  Stage 1 if GFR value is ≥90; Stage 2 if 60 ≤ GFR < 90; Stage 3A if 45 ≤ GFR < 60; Stage 3B if 30 ≤ GFR < 45; Stage 4 if 15 ≤ GFR < 30; Stage 5 if GFR < 15.
  Stage 1 means kidney function is normal. Stage 2 indicates mildly reduced kidney function, pointing to kidney disease. Stages 3A abd 3B indicate moderately reduced kidney function. Stage 4 indicates severely reduced kidney function. Stage 5 indicates very severe or end stage kidney failure.
Time Frame: Week 52, Week 104, and Week 156
Population: Intent-to-treat population with available data at Weeks 52, 104 and 156
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 4 | 3 | 7
Participants
  Week 52 | 0 | 1 | 0
  Week 104: number analyzed (Participants) | 3 | 2 | 7
  Week 104 | 0 | 0 | 0
  Week 156: number analyzed (Participants) | 3 | 2 | 7
  Week 156 | 0 | 0 | 0

6. Secondary Outcome: Mean Calculated eGFR Using MDRD 4 Variable Model
Description: The estimated Glomerular Filtration Rate (eGFR) was calculated using the Modification of Diet in Renal Disease equation (MDRD). A score of ≥90 means kidney function is normal. A score between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease. Scores between 30 and 59 indicates moderately reduced kidney function. Scores between 15 and 29 indicate severely reduced kidney function. Scores below 15 indicate very severe or endstage kidney failure.
Time Frame: Week 52, Week 104, and Week 156
Population: Intent-to-treat population with available data at Weeks 52, 104 and 156
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 4 | 3 | 7
mL/min/1.73m^2
  Week 52 | 52.4 (8.3) | 47.8 (22.3) | 55.7 (11.0)
  Week 104: number analyzed (Participants) | 3 | 2 | 7
  Week 104 | 54.2 (13.1) | 69.3 (27.3) | 60.4 (16.8)
  Week 156: number analyzed (Participants) | 3 | 2 | 7
  Week 156 | 49.0 (16.3) | 65.5 (20.2) | 61.5 (13.9)

7. Secondary Outcome: The Slope of eGFR by CKD-EPI Over Time Based on Serum Creatinine
Description: The estimated Glomerular Filtration Rate (eGFR) was calculated using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI). A score of ≥90 means kidney function is normal. A score between 60 and 89 indicates mildly reduced kidney function, pointing to kidney disease. Scores between 30 and 59 indicates moderately reduced kidney function. Scores between 15 and 29 indicate severely reduced kidney function. Scores below 15 indicate very severe or endstage kidney failure. An estimate of the slope, or change over time, in eGFR was produced using standard statistical linear modeling procedures. The estimate was then re-scaled so that it can be interpreted as a change in eGFR per month. Positive numbers indicate increasing kidney function. Larger numbers indicate greater change in kidney function.
Time Frame: Week 52, Week 104, and Week 156
Population: Intent-to-treat with available data
Measure: Mean (Standard Deviation); unit: Change in eGFR (mL/min/1.73m^2) by month
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 4 | 7
Change in eGFR (mL/min/1.73m^2) by month
  Week 52 | 1.29 (1.85) | 0.62 (0.99) | 1.07 (1.16)
  Week 104 | 1.27 (1.86) | 0.62 (1.18) | 0.68 (0.83)
  Week 156 | 1.33 (1.82) | 0.69 (1.14) | 0.48 (0.48)

8. Secondary Outcome: Count of Participants With Delayed Graft Function Post-Transplant
Description: Delayed graft function is defined as dialysis in the first week on one or more occasions for any indication other than the treatment of acute hyperkalemia in the setting of otherwise acceptable renal function
Time Frame: Any time within the first week post-transplant
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Participants | 0 | 2 | 0

9. Secondary Outcome: An Increase of One or More Grades of CAN/IFTA When Comparing the Implantation and Subsequent Protocol Biopsies
Description: CAN/IFTA grades reflect the severity of interstitial fibrosis and tubular atrophy present in the tissue obtained during a kidney biopsy. Higher grades indicate greater severity in interstitial fibrosis and tubular atrophy present the kidney biopsy tissue. The aim of this measure was to compare central lab reviewed pre-implantation biopsies to post-transplant biopsies, as pre-specified per protocol; however, the central lab had an inadequate set of biopsies to proceed with evaluation.
Time Frame: Week 52, Week 104, and Week 156
Population: There was an insufficient number of biopsies collected for the summarized data to be reliable.
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Count of Participants With CAN/IFTA Grade I, II or III at Any Time Post-transplant
Description: CAN/IFTA grades were determined per local pathology interpretations of biopsy tissue. These grades reflect the severity of interstitial fibrosis and tubular atrophy present in the tissue obtained during a kidney biopsy. Higher grades indicate greater severity in interstitial fibrosis and tubular atrophy present the kidney biopsy tissue.
Time Frame: Transplantation through last study visit (up to week 156)
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Participants | 1 | 3 | 5

11. Secondary Outcome: Count of Participants With Acute Cellular Rejection Grade Equal to or Greater Than IA, by the Banff 2007 Criteria
Description: Acute cellular rejection is when lesions at the site of the graft characteristically are infiltrated with large numbers of lymphocytes and macrophages that cause tissue damage. Acute cellular rejection for this endpoint is defined as a grade ≥ IA by Banff 2007 criteria.
Time Frame: Transplantation through last study visit (up to week 156)
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Participants | 0 | 2 | 4

12. Secondary Outcome: Count of Participants by Severity of First Acute Cellular Rejection by Wk 52
Description: Acute cellular rejection is when lesions at the site of the graft characteristically are infiltrated with large numbers of lymphocytes and macrophages that cause tissue damage. Acute cellular rejection for this endpoint is defined as a grade ≥ IA by Banff 2007 criteria. Severity is graded as IA, IB, IIA, IIB, or III, with IA being the mildest form of cellular rejection and III being the most severe form of cellular rejection. Originally, this endpoint was worded as "The severity of first and highest acute cellular rejection within the first 52 weeks." But since the highest grade for each subject coincided with the first ACR episode for each subject, only a summary of severity of the first episode is presented here.
Time Frame: Transplantation through Week 52
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Participants
  Grade IA | 0 | 1 | 1
  Grade IB | 0 | 0 | 0
  Grade IIA | 0 | 0 | 2
  Grade IIB | 0 | 1 | 1
  Grade III | 0 | 0 | 0

13. Secondary Outcome: Count of Participants With Antibody Mediated Rejection
Description: Antibody mediated rejection (AMR) is defined as diffusely positive staining for C4d, presence of circulating anti-donor antibodies and morphologic evidence of acute tissue injury.
Time Frame: Transplantation through last study visit (up to week 156)
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Participants | 0 | 1 | 0

14. Secondary Outcome: Type of Treatment of Rejection
Description: Upon having a biopsy performed, persons often receive treatment for rejection based on the results of the biopsy, which may or may not have shown signs of rejection. Details of biopsy findings and corresponding treatment are presented here for each instance of treatment for rejection. Acronyms and abbreviations are defined below.
  ACR=Acute Cellular Rejection ATG=Anti-thymocyte globulin therapy Chr. AMR=Chronic Antibody Mediated Rejection Gd.=Grade IFTA=Interstitial Fibrosis and Tubular Atrophy IVIG=Intravenous Immunoglobulin therapy.
  Only 'for cause' biopsies were performed post-transplant; thus, it is possible for a participant to be included in the analysis population and not have a biopsy for this outcome measure.
Time Frame: Transplantation through last study visit (up to week 156)
Population: Intent-to-treat
Measure: Number; unit: Biopsy
Units Other Than Participants: Biopsies
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Number analyzed (Biopsies) | 5 | 10 | 10
Biopsy
  Borderline rejection; IVIG and plasmapheresis | 1 | 0 | 0
  ACR Gd. IA + Chr. AMR + IFTA Gd. I; Pulse Steroids | 0 | 1 | 0
  ACR Gd. IA + IFTA Gd. II; Pulse Steroids | 0 | 1 | 0
  ACR Gd. IIB; ATG and Pulse Steroids | 0 | 1 | 0
  Borderline + IFTA Gd. I; with Pulse Steroids | 0 | 0 | 1
  ACR Gd. IA + IFTA Gd. I; Pulse Steroids | 0 | 0 | 1
  ACR Gd. IIA; Pulse Steroids | 0 | 0 | 1
  ACR Gd. IIA + IFTA Gd. I; ATG and Pulse Steroids | 0 | 0 | 2
  ACR Gd. IIB + IFTA Gd. I; ATG and Pulse Steroids | 0 | 0 | 1

15. Secondary Outcome: Count of Participants With de Novo Anti-donor HLA Antibodies at Wk 52
Description: The presence of antibodies reactive to Histocompatibility Antigen (HLA) molecules expressed on the renal allograft have been associated with both acute and chronic injury to the transplanted kidney. The development of de novo anti- donor HLA antibodies may mean a person is more likely to reject the graft.
Time Frame: Week 52
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Participants | 0 | 0 | 0

16. Secondary Outcome: Count of Participants With Either New Onset Diabetes After Transplant (NODAT) or Impaired Fasting Glucose (IFG) at Wk 52 Based on Criteria Specified by the ADA and WHO
Description: New onset diabetes is the development of diabetes post-kidney transplant. It was identified by the clinical sites caring for each participant and reported directly in the clinical database. Impaired fasting glucose (IFG) is a determination made by referencing glucose measurements obtained from a standard chemistry panel. Any fasting glucose measure that is between 110 and 125 mg/dL is classified as IFG.
  Acronyms: American Diabetes Association (ADA); World Health Organization (WHO).
Time Frame: Week 52
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Participants
  New onset diabetes during first 52 weeks | 0 | 0 | 0
  Impaired fasting glucose at week 52: number analyzed (Participants) | 4 | 2 | 6
  Impaired fasting glucose at week 52 | 1 | 0 | 0

17. Secondary Outcome: Count of Participants With Treated Diabetes Between Day 14 and Wk 52
Description: Treated diabetes is defined as the receipt of oral medication or insulin for >14 days between 14 days and 52 weeks post-transplant
Time Frame: Day 14 to Week 52
Population: Intent-to-treat with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 4 | 3 | 7
Participants | 1 | 0 | 1

18. Secondary Outcome: HbA1c Measured at Days 28 & 84, and Weeks 24, 36, 52, 72, 104 and 156
Description: Hemoglobin A1c (HbA1c) measures the average blood glucose levels over 8-12 weeks, thus acting as a useful long-term gauge of blood glucose control. A value below 6.0% reflects normal levels, 6.0% to 6.4% reflects prediabetes, and a value of ≥ 6.5% reflects diabetes.
Time Frame: Day 28, Day 84, Week 24, Week 36, Week 52, Week 72, Week 104, Week 156
Population: Intent-to-treat with available data
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 4 | 7
percent
  Day 28: number analyzed (Participants) | 6 | 4 | 6
  Day 28 | 5.3 (1.1) | 5.1 (0.5) | 5.8 (0.2)
  Day 84: number analyzed (Participants) | 5 | 4 | 7
  Day 84 | 5.7 (1.4) | 5.0 (0.6) | 5.9 (0.8)
  Week 24: number analyzed (Participants) | 4 | 3 | 6
  Week 24 | 6.9 (1.8) | 5.1 (0.3) | 6.5 (1.0)
  Week 36: number analyzed (Participants) | 2 | 2 | 4
  Week 36 | 6.7 (1.5) | 5.3 (0.4) | 7.2 (2.6)
  Week 52: number analyzed (Participants) | 3 | 2 | 1
  Week 52 | 7.0 (2.9) | 4.8 (0.7) | 7.6
  Week 72: number analyzed (Participants) | 0 | 0 | 1
  Week 72 |  |  | 8.1
  Week 104: number analyzed (Participants) | 2 | 2 | 5
  Week 104 | 5.7 (0.4) | 5.2 (0.1) | 6.6 (1.8)
  Week 156: number analyzed (Participants) | 2 | 2 | 6
  Week 156 | 5.6 (0.1) | 5.2 (0.1) | 7.8 (2.5)

19. Secondary Outcome: Standardized Blood Pressure Measurement at Wk 52
Description: A blood pressure measurement consists of two numbers: the systolic and diastolic pressures. Systolic pressure measures the pressure in blood vessels when the heart beats. Diastolic pressure measures the pressure in blood vessels between beats of the heart. Systolic measures of <120 and diastolic measures of <80 are considered normal. Systolic measures of 120-139 and diastolic measures of 80-89 are considered at risk (or pre-hypertension). Systolic measures of ≥140 and diastolic measures of ≥90 are considered high.
Time Frame: Week 52
Population: Intent-to-treat with available data at Week 52
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 4 | 3 | 7
mmHg
  Systolic Blood Pressure at Week 52 | 147.5 (18.7) | 146.7 (5.1) | 139.9 (18.1)
  Diastolic Blood Pressure at Week 52 | 80.8 (12.8) | 92.7 (9.8) | 79.3 (8.5)

20. Secondary Outcome: Count of Participants With Use of Anti-hypertensive Medications at Wk 52
Description: Anti-hypertensive medications are a class of drugs that are used to treat hypertension. The medications seek to prevent the complications of high blood pressure, such as stoke and myocardial infarction.
Time Frame: Week 52
Population: Intent-to-treat with available data at Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 4 | 3 | 7
Participants | 3 | 3 | 7

21. Secondary Outcome: Fasting Lipid Profile (Total Cholesterol, Non-HDL Cholesterol, LDL, HDL, and Triglyceride) at Baseline and Wks 24, 52, 104 and 156
Description: A fasting lipid profiles measures total cholesterol, LDL cholesterol, HDL cholesterol, and triglyceride levels. These measurements are used in assessing one's risk of cardiovascular disease. Target ranges for each of these measures are detailed below.
  Total cholesterol: 75-169 mg/dL if age ≤ 20; 100-199 mg/dL if age ≥ 21; high values indicate risk of cardiovascular disease
  LDL cholesterol: <70 mg/dL for people with documented cardiovascular disease or metabolic syndrome; <100 mg/dL for people considered high risk for cardiovascular disease; <130 mg/dL for people considered low risk for cardiovascular disease; high values indicate risk of cardiovascular disease
  HDL cholesterol: 40mg/dL and higher; high values indicate reduced risk of cardiovascular disease
  Non-HDL cholesterol: 30 mg/dL above the target value for LDL cholesterol; high values indicate risk of cardiovascular disease
  Triglycerides: <150 mg/dL; high values indicate risk of cardiovascular disease
Time Frame: Baseline, Week 24, Week 52, Week 104, Week 156
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
mg/dL
  Tot. Chol. Baseline | 141.2 (28.8) | 160.2 (37.8) | 165.6 (37.4)
  Tot. Chol. W24: number analyzed (Participants) | 5 | 3 | 7
  Tot. Chol. W24 | 171.6 (44.0) | 159.0 (11.1) | 185.6 (40.1)
  Tot. Chol. W52: number analyzed (Participants) | 4 | 1 | 2
  Tot. Chol. W52 | 156.0 (30.7) | 187.0 | 157.5 (53.0)
  Tot. Chol. W104: number analyzed (Participants) | 2 | 2 | 5
  Tot. Chol. W104 | 170.5 (2.1) | 142.5 (3.5) | 189.0 (49.9)
  Tot. Chol. W156: number analyzed (Participants) | 2 | 2 | 6
  Tot. Chol. W156 | 183.5 (3.5) | 133.5 (7.8) | 181.7 (60.6)
  Non-HDL Baseline | 108.2 (22.0) | 118.8 (19.0) | 122.3 (44.9)
  Non-HDL W24: number analyzed (Participants) | 5 | 3 | 7
  Non-HDL W24 | 128.0 (38.0) | 129.3 (10.0) | 129.0 (35.3)
  Non-HDL W52: number analyzed (Participants) | 4 | 1 | 1
  Non-HDL W52 | 117.5 (23.4) | 151.0 | 61.0
  Non-HDL W104: number analyzed (Participants) | 2 | 2 | 5
  Non-HDL W104 | 129.5 (0.7) | 110.5 (3.5) | 135.6 (42.4)
  Non-HDL W156: number analyzed (Participants) | 2 | 2 | 6
  Non-HDL W156 | 138.5 (2.1) | 102.5 (2.1) | 136.0 (58.0)
  LDL Baseline | 76.7 (22.0) | 86.6 (29.8) | 83.4 (41.4)
  LDL W24: number analyzed (Participants) | 5 | 3 | 7
  LDL W24 | 76.7 (22.0) | 86.6 (29.8) | 83.4 (41.4)
  LDL W52: number analyzed (Participants) | 4 | 1 | 1
  LDL W52 | 69.5 (38.0) | 114.0 | 49.0
  LDL W104: number analyzed (Participants) | 2 | 2 | 5
  LDL W104 | 100.5 (0.7) | 58.0 (18.4) | 101.4 (42.3)
  LDL W156: number analyzed (Participants) | 2 | 2 | 6
  LDL W156 | 116.0 (2.8) | 55.5 (19.1) | 106.0 (46.3)
  HDL Baseline | 33.0 (10.4) | 41.3 (22.8) | 43.3 (10.7)
  HDL W24: number analyzed (Participants) | 5 | 3 | 7
  HDL W24 | 43.6 (8.2) | 29.7 (2.1) | 56.6 (19.6)
  HDL W52: number analyzed (Participants) | 4 | 1 | 1
  HDL W52 | 38.5 (12.3) | 36.0 | 59.0
  HDL W104: number analyzed (Participants) | 2 | 2 | 5
  HDL W104 | 41.0 (2.8) | 32.0 (7.1) | 53.4 (16.6)
  HDL W156: number analyzed (Participants) | 2 | 2 | 6
  HDL W156 | 45.0 (1.4) | 31.0 (5.7) | 45.7 (14.6)
  Triglyc. Baseline | 158.7 (92.4) | 307.8 (350.1) | 206.9 (148.5)
  Triglyc. W24: number analyzed (Participants) | 5 | 3 | 7
  Triglyc. W24 | 161.0 (53.9) | 249.7 (172.4) | 115.9 (68.1)
  Triglyc. W52: number analyzed (Participants) | 4 | 1 | 1
  Triglyc. W52 | 319.3 (294.0) | 187.0 | 58.0
  Triglyc. W104: number analyzed (Participants) | 2 | 2 | 5
  Triglyc. W104 | 146.0 (1.4) | 220.0 (168.3) | 172.8 (130.0)
  Triglyc. W156: number analyzed (Participants) | 2 | 2 | 6
  Triglyc. W156 | 115.0 (4.2) | 228.0 (93.3) | 156.5 (75.6)

22. Secondary Outcome: Count of Participants With Use of Lipid Lowering Medications at Baseline and Wks 24, 52, 104 and 156
Description: Lipid lowering medications are used in the treatment of high levels of fats (lipids), such as cholesterol in blood
Time Frame: Baseline, Week 24, Week 52, Week 104, Week 156
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Participants
  Baseline | 5 | 1 | 2
  Week 24: number analyzed (Participants) | 6 | 4 | 7
  Week 24 | 4 | 1 | 2
  Week 52: number analyzed (Participants) | 4 | 3 | 7
  Week 52 | 3 | 1 | 2
  Week 104: number analyzed (Participants) | 4 | 3 | 7
  Week 104 | 3 | 1 | 3
  Week 156: number analyzed (Participants) | 4 | 2 | 7
  Week 156 | 3 | 1 | 3

23. Secondary Outcome: Total Daily Prescribed Pill Number at Days 28 and 84, and Wks 24, 36, 52, 72, 104 and 156
Description: This is a measure of the total number of pills a participant was prescribed on a given day
Time Frame: Day 28, Day 84, Week 24, Week 36, Week 52, Week 72, Week 104, Week 156
Population: Intent-to-treat with available data
Measure: Mean (Standard Deviation); unit: Number of pills
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 4 | 7
Number of pills
  Day 28 | 28.8 (12.3) | 15.8 (6.3) | 27.3 (7.6)
  Day 84 | 22.2 (6.6) | 13.5 (4.4) | 21.3 (7.5)
  Week 24: number analyzed (Participants) | 5 | 3 | 7
  Week 24 | 14.8 (3.8) | 8.3 (4.0) | 16.6 (5.7)
  Week 36: number analyzed (Participants) | 3 | 3 | 7
  Week 36 | 13.0 (2.0) | 14.0 (1.0) | 17.0 (5.1)
  Week 52: number analyzed (Participants) | 4 | 3 | 6
  Week 52 | 14.6 (5.0) | 14.3 (1.5) | 17.8 (3.5)
  Week 72: number analyzed (Participants) | 0 | 0 | 4
  Week 72 |  |  | 16.0 (4.4)
  Week 104: number analyzed (Participants) | 4 | 2 | 6
  Week 104 | 15.3 (5.7) | 15.5 (2.1) | 14.8 (5.3)
  Week 156: number analyzed (Participants) | 4 | 2 | 7
  Week 156 | 14.0 (6.2) | 15.0 (1.4) | 12.7 (6.2)

24. Secondary Outcome: Number of Events of Death or Graft Loss
Description: This measure counts deaths and graft loss occurring at any point post transplantation. Graft loss is defined as need for dialysis for greater than 30 days duration, allograft nephrectomy, or retransplantation.
Time Frame: Transplantation through last study visit (up to week 156)
Population: Intent-to-treat
Measure: Number; unit: Events
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Events | 2 | 3 | 0

25. Secondary Outcome: Count of Participants With Rejection
Description: The number of participants who were treated by their local physician for any type of rejection including, but not limited to cellular rejection and antibody- mediated rejection of the transplanted kidney regardless of the presence of a biopsy.
Time Frame: Transplantation through last study visit (up to week 156)
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Participants | 1 | 3 | 5

26. Secondary Outcome: Number of All Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Adverse events were collected systematically from enrollment through last study visit. Displayed below are counts of all adverse events per treatment group (including both serious and non-serious adverse events). Separately counts of all adverse events determined to be serious are displayed per treatment group. More detail about adverse events for this trial is displayed in the 'Adverse Event' section.
Time Frame: Enrollment through last study visit (up to week 156)
Population: Intent-to-treat
Measure: Number; unit: Events
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Events
  All Adverse Events | 21 | 25 | 40
  Serious Adverse Events | 6 | 11 | 7

27. Secondary Outcome: Count of Participants With Infections Requiring Hospitalization or Systemic Therapy Reported as Serious Adverse Events
Description: Infections of certain types (i.e., excluding those identified in the protocol as occurring commonly in this study population) were required to be reported as a serious adverse event if they required either inpatient hospitalization of prolongation of a current hospitalization.
Time Frame: Transplantation through last study visit (up to week 156)
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Participants | 2 | 2 | 1

28. Secondary Outcome: Count of Participants With BKV and CMV Viremia (Local Center Monitoring) Reported as Adverse Events
Description: Viral infections following renal transplantation is significant source of recipient morbidity and mortality, and a significant cause of allograft dysfunction and loss. Specific viruses were monitored during this study using participant blood samples.
  Acronyms: BK Polyoma Virus (BKV); Cytomegalovirus (CMV).
Time Frame: Transplantation through last study visit (up to week 156)
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Participants
  BKV | 0 | 0 | 2
  CMV | 1 | 0 | 0

29. Secondary Outcome: Count of Participants With EBV Infection as Reported on the Case Report Form as Adverse Events
Description: Viral infections following renal transplantation is a significant source of recipient morbidity and mortality, and a significant cause of allograft dysfunction and loss. Specific viruses were monitored during this study using participant blood samples.
  Acronym: Epstein-Barr virus (EBV)
Time Frame: Transplantation through last study visit (up to week 156)
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Participants | 0 | 0 | 0

30. Secondary Outcome: Count of Participants With Fever > 39 Degrees Celsius and Blood Pressure < 90mm Hg Within 24 Hours of Onset of Transplant Procedure
Description: Temperature of >39 degrees Celsius would be an indication of fever most often in response to an infection or illness. Systolic blood pressure <90mm Hg would be an indication of low blood pressure.
Time Frame: 24 hours after transplantation
Population: Intent-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
Number analyzed (Participants) | 6 | 6 | 7
Participants
  Fever >39 degrees | 0 | 0 | 0
  Systolic BP <90 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Enrollment through study completion, up to 3 years
Arm/Group | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus | Induction: Alemtuzumab, Maintenance: MMF + Belatacept | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac
All-Cause Mortality (participants affected / at risk) | 1/6 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/6 | 5/6 | 5/7
Other Adverse Events (participants affected / at risk) | 6/6 | 4/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus (N=6) | Induction: Alemtuzumab, Maintenance: MMF + Belatacept (N=6) | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac (N=7)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 1 (1) | 3 (3)
Arteriovenous graft site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endocarditis staphylococcal (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Renal vein thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction: Alemtuzumab, Maintenance: MMF + Tacrolimus (N=6) | Induction: Alemtuzumab, Maintenance: MMF + Belatacept (N=6) | Induction: Basiliximab, Maintenance: MMF + Belatacept + Tac (N=7)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (5)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Type IV hypersensitivity reaction (Immune system disorders) | 0 (0) | 1 (1) | 2 (2)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (4)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 2 (5)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haematocrit increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Polyomavirus test positive (Investigations) | 0 (0) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Renal artery thrombosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment of 210 participants was planned, but study was stopped after 19 participants enrolled due to safety concerns and change in alemtuzumab availability. Enrolled participants continued follow-up after enrollment ended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No